CLINICAL TRIAL: NCT02343055
Title: Collaborative Self-Management Patient Education Will Improve Health Outcomes in COPD
Brief Title: COPE With COPD Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Pfizer (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00000941
Record Dates: First submitted 2014-10-22; First posted 2015-01-21 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2015-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Case Management and Self-Management Education (Experimental): A Certified Respiratory Educator (CRE) will obtain a detailed COPD history, provide general and self-management education, and confirm a management plan with the primary care physician. Specific elements of evidence-based management are targetted for intervention. Subjects will return for a follow-up visit in-person with the interdisciplinary care team including a CRE to review their health status including COPD symptoms, exacerbation diary, symptoms, MRC scale, etc as a minimum at 3 and 12 months. Telephone follow up will occur at a minimum at 6 and 9 months.
  Interventions: Other: Case Management and Self-Management Education
- Usual Care (Placebo Comparator): A Certified Respiratory Educator (CRE) will meet with subjects to obtain a detailed COPD history and do a breathing test. Subjects will receive COPD care as usually provided by their physician.
  Interventions: Other: Case Management and Self-Management Education

INTERVENTIONS:
Other: Case Management and Self-Management Education — A Certified Respiratory Educator (CRE) will obtain a detailed COPD history, provide general and self-management education, and confirm a management plan with the primary care physician. Specific elements of evidence-based management are targetted for intervention. Subjects will return for a follow-up visit in-person with the interdisciplinary care team including a CRE to review their health status including COPD symptoms, exacerbation diary, symptoms, MRC scale, etc as a minimum at 3 and 12 months. Telephone follow up will occur at a minimum at 6 and 9 months.

SUMMARY:
The overall objective of this study is to evaluate a collaborative self-management intervention in patients with moderate to severe COPD in a primary care population. To achieve this objective the investigators developed a diagnostic and treatment pathway for the management of COPD in primary care that is based on national guidelines and focused on patient self-management.

.

ELIGIBILITY:
Inclusion Criteria:

* Current or Ex-smokers
* 40 years of age or over
* Minimum 10 pack year smoking history
* Post-bronchodilator FEV1 of 70% or less (4 puffs of Salbutamol) and Forced Expiratory Volume at 1sec to Forced Vital Capacity (FEV1/FVC) ratio 70% or less
* A history of two exacerbations (involving treatment and/or visit to a health care practitioner) in the past 3 years OR 1 exacerbation in the past year
* Provides informed consent

Exclusion Criteria:

* COPD exacerbation in the past 4 weeks
* Diagnosis of asthma prior to the age of 40 years
* Co-existing illness that could interfere with study results (ie. Congestive Heart Failure with exacerbation of symptoms)
* Scheduled for COPD rehabilitation
* A terminal illness

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2011-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) | 1 Year
  COPD related quality of life measure in primary care.

SECONDARY OUTCOMES:
Health Care Utilization for Emergency Department visits proportion and rate per year | 1 year
  The proportion of subjects that utilized the Emergency for a COPD exacerbation
Health Care Utilization for Hospital Admission proportion and rate per year | 1 year
  The proportion of subjects that were admitted to hospital for a COPD exacerbation An exacerbation is defined as an increase in or the onset of more than one respiratory symptom (cough, sputum, sputum purulence, wheezing, or dyspnea) lasting 3 days or more and requiring treatment with an antibiotic or a systemic corticosteroid. Respiratory status had to return to baseline for at least 72 hours before another exacerbation would be counted.
Severe Exacerbation proportion and rate per year | 1 year
  The proportion of subjects experiencing one or more exacerbations in the study interval. An exacerbation diary will be completed for each event.

OTHER OUTCOMES:
Quality of Life | 1 year
  Improvement of Quality of Life using the CAT score(COPD Assessment Test)
Improvement in Knowledge of COPD and confidence in self-management | 1 year
  Improvement in Bristol COPD Knowledge Questionnaire and patient self report
Process of Care | 1 year
  Process of care: have written action plan, used action plan, advised to quit smoking, offered pharmacologic help with quitting, quit smoking, current packs/day, diagnosis confirmed by spirometry, vaccination rates, instructed on inhaler technique, vaccination rates
Dyspnea Improvement | 1 year
  Change in dyspnea using the modified MRC questionnaire - Medical Research Council (MRC).
Disease control | 1 year
  Disease control using the Clinical COPD questionnaire (CCQ)
Symptom Profile | 1 year
  Change in Symptom profile (cough, wheeze, sputum production)
Forced Expiratory Volume at 1sec (FEV1) % predicted | 1 year
  FEV1
Proportion of Patients on therapy appropriate to their stage of disease | 1 year
  Evaluate medication prescribed related to stage of disease

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Licskai, Principal Investigator — Lawson Health Research Institution
Locations (4):
- Canada (4):
  - Amherstburg FHT, Amherstburg, Ontario
  - Chatham-Kent FHT, Chatham, Ontario
  - Harrow FHT, Harrow, Ontario
  - Leamington FHT, Leamington, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrone M, Masciantonio MG, Malus N, Stitt L, O'Callahan T, Roberts Z, Johnson L, Samson J, Durocher L, Ferrari M, Reilly M, Griffiths K, Licskai CJ; Primary Care Innovation Collaborative. The impact of integrated disease management in high-risk COPD patients in primary care. NPJ Prim Care Respir Med. 2019 Mar 28;29(1):8. doi: 10.1038/s41533-019-0119-9. PMID 30923313